CLINICAL TRIAL: NCT05626400
Title: Clinical Study of Senl-T7 CAR T Cells in the Treatment of Relapsed and Refractory CD7+ Acute T Lymphoblastic Leukemia and T Lymphoblastic Lymphoma
Brief Title: Clinical Study of Senl-T7 CAR T Cells in the Treatment of Relapsed and Refractory CD7+ Acute T-ALL/T-LBL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Senl-T7 CAR for T-ALL/T-LBL
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-08

CONDITIONS: T-cell Acute Lymphoblastic Leukemia/Lymphoma
Keywords: T-ALL; T-LBL; CD7; CAR-T
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD-7 CART (Experimental): Patients will be treated with CD7 CAR-T cells
  Interventions: Biological: Senl-T7

INTERVENTIONS:
Biological: Senl-T7 — Patients will be treated with CD7 CAR-T cells

SUMMARY:
This is an open, prospective, dose-escalation clinical study to evaluate the safety and efficacy of Senl-T7 in patients with relapsed or refractory CD7+ acute T lymphoblastic leukemia or T lymphoblastic lymphoma.Meanwhile, PK/PD indexes of Senl-T7 were collected.

DETAILED DESCRIPTION:
The CARs consist of an anti-CD7 single-chain variable fragment（scFv）, a portion of the human CD137（4-1BB） molecule, and the intracellular component of the human CD3ζ molecule. Prior to CAR-T cell infusion, the patients will be subjected to preconditioning treatment. After CAR-T cell infusion, the patients will be evaluated for adverse reactions and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsed/refractory T-cell lymphoblastic leukemia or T-cell lymphoblastic lymphoma: Induction therapy failed to achieve a complete remission of minor residual negative; Recurrence: after complete remission, any tumor load in the peripheral blood or bone marrow was 5%, or slightly residual positive, or new extramedullary lesions occurred；
2. CD7 expression in tumor cells was detected by flow cytometry；
3. Life expectancy greater than 12 weeks；
4. KPS or Lansky score≥60;
5. HGB≥70g/L (can be transfused);
6. 2-70 years old;
7. Oxygen saturation of blood#90%#;
8. HGB≥70g/L（blood transfusion allowed）;
9. Total bilirubin (TBil)≤3 × upper limit normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal;
10. Informed consent explained to, understood by and signed by patient/ guardian.

Exclusion Criteria:

1. Any of the following cardiac criteria: Atrial fibrillation/flutter; Myocardial infarction within the last 12 months; Prolonged QT syndrome or secondary prolonged QT, per investigator discretion. Cardiac echocardiography with LVSF (left ventricular shortening fraction)<30% or LVEF(left ventricular ejection fraction)<50%; or clinically significant pericardial effusion. Cardiac dysfunction NYHA(New York Heart Association) III or IV (Confirmation of absence of these conditions on echocardiogram within 12 months of treatment);
2. Has an active GvHD;
3. Has a history of severe pulmonary function damaging;
4. With other tumors which is/are in advanced malignant and has/have systemic metastasis;
5. Severe or persistent infection that cannot be effectively controlled;
6. Merging severe autoimmune diseases or immunodeficiency disease;
7. Patients with active hepatitis B or hepatitis C([HBVDNA+]or [HCVRNA+]);
8. Patients with HIV infection or syphilis infection;
9. Has a history of serious allergies on Biological products (including antibiotics);
10. Clinically significant viral infection or uncontrolled viral reactivation of EBV(Epstein-Barr virus), CMV(cytomegalovirus), ADV(adenovirus), BKvirus, or HHV(human herpesvirus)-6;
11. Presence of symptomatic disorders of the central nervous system, which include but not limited to uncontrolled epilepsy, cerebrovascular ischemia/hemorrhage, dementia, and cerebellar disease, etc.;
12. Have received transplant treatment for less than 6 months in prior to enrollment;
13. Being pregnant and lactating or having pregnancy within 12 months;
14. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after CD7 CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Remission Rate | 3 months post CAR-T cells infusion
  To obsere the efficacy of CAR-T cells after infusion, complete remission (CR), complete remission with incomplete recovery of blood cells (CRi), minimal tumor residual positive(MRD+) or negative (MRD-) CR/CRi, disease recurrence or progression (PD) will be used for evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei yanda Hospital, Beijingcun, Hebei, China